CLINICAL TRIAL: NCT03067090
Title: Prospective Study of Aquamid Reconstruction in Patients With Osteoarthritis of the Knee
Brief Title: Aquamid Reconstruction for Osteoarthritis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: A2 Reumatologi Og Idrætsmedicin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2-001
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-articular Aquamid Reconstruction (Experimental): Intra-articular injection of 3 ml aquamid reconstruction (AR) to the knee. A second injection of 3 ml will take place after 1 month (+/- 2 weeks).
  Interventions: Device: Aquamid Reconstruction

INTERVENTIONS:
Device: Aquamid Reconstruction — AR contains 2.5% polyacrylamide and 97.5% non-pyrogenic water, with a unique molecular structure that allows the normal water exchange with the surrounding tissue without losing shape or effect. AR is biocompatible, non-biodegradable, stable and sterile.
  The gel is provided in a sterile, pre-filled 1 ml sealed syringe. The gel is intended to be injected intra-articularly with a sterile 21G x 2 inch (0.8 x 50 mm) needle.

SUMMARY:
Osteoarthritis (OA) causes degradation and deformities of joints, including knees, hips, hands, and feet. Approximately more than 55% of populations above 45 years and more than 70% of population above 70 years will develop OA in at least one joint. The symptoms are dominated by pain but also stiffness and swelling occur. There is currently no cure for OA, and the ultimate treatment is joint replacement surgery. However, there is an unmet need to identify other treatment options that may delay or avoid surgery.

Aquamid Reconstruction (AR) is a polyacrylamide hydrogel (PAAG) which is a non-degradable, highly visco-elastic synthetic gel, which is atoxic with durable effect and tissue-compatibility and well tolerated by mammal tissue by allowing in vivo vessel and fibrous in-growth. Experimental studies supported by histopathological observations have shown that AR exerts its effect via integration over time within the soft tissues, through a combination of vessel in-growth and molecular water exchange. Intra-articular injection of AR is expected to provide permanent pain relief and improve the functional ability through a cushioning or padding effect on the joint and thereby reduce symptoms and improve patients' quality of life.

The purpose of this study is to obtain information of the safety and effectiveness of AR in patients with OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* WOMAC pain score >/= 5
* Kellgren and Lawrence radiographic scoring >/= 1
* Signed informed consent form

Exclusion Criteria:

* Other diseases affecting the joints such as rheumatoid arthritis
* Actual or recurrent infections requiring intravenous antibiotic treatment within the last 30 days or oral antibiotic treatment within the last 14 days before inclusion
* Less than 12 weeks since injection of HA or corticosteroids in study-knee joint before treatment
* Pregnancy or lactation
* Not able to comply with the requirements of the study
* Previous alloplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the pain subscore of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 6 months
  The WOMAC is a patient reported questionnaire that is easy to use and evaluates three domains; pain (five questions), stiffness (two questions) and physical function (17 questions), each weighted on a similar computation. The WOMAC Index is sensitive to change and is valid for elderly subjects with knee OA.

SECONDARY OUTCOMES:
Change from baseline in all subscores of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 3, 6 and 12 months
  The WOMAC is a patient reported questionnaire that is easy to use and evaluates three domains; pain (five questions), stiffness (two questions) and physical function (17 questions), each weighted on a similar computation. The WOMAC Index is sensitive to change and is valid for elderly subjects with knee OA.
Participants' percieved effect | 1, 3, 6, and 12 months
  Participants will be surveyed about the current state of the treated knee. Predefined answers are: Worsened; No change; Improved; Cured.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hartkopp, Principal Investigator — A2 Reumatologi of idrætsmedicin
Locations (1):
- A2 reumatologi og idrætsmedicin, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided